CLINICAL TRIAL: NCT03697798
Title: Immunological Effects of an Acellular Pertussis Booster Vaccination in Children, Young Adults and Elderly With Different Immunisation Background. An International Study in Finland, the Netherlands and the United Kingdom
Brief Title: A Study Exploring Whooping Cough Protection in Children and Adults
Acronym: BERT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government); University of Turku (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OVG 2016/05
Record Dates: First submitted 2018-04-23; First posted 2018-10-05 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pertussis
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Children aged between 7-10 years of age (Active Comparator): Healthy children from 7 up to 10 years of age, determined by date of birth (dd/mm/yyyy), at the time of the first visit. Male + female, approximately equally distributed, n = 36 in each country. They will receive Boostrix®-IPV combination vaccine.
  Interventions: Biological: Boostrix®-IPV combination vaccine
- Children aged between 11-15 years of age (Active Comparator): Healthy children from 11 up to 15 years of age, determined by date of birth (dd/mm/yyyy), at the time of the first visit. Male + female, approximately equally distributed, n = 36 in each country aiming for comparable numbers of participants with aP vs wP vaccination background. They will receive Boostrix®-IPV combination vaccine.
  Interventions: Biological: Boostrix®-IPV combination vaccine
- Adults aged between 20-34 years of age (Active Comparator): Healthy young adults from 20 up to 34 years of age, determined by date of birth (dd/mm/yyyy), at the time of the first visit. Male + female, approximately equally distributed, n = 25 in each country. They will receive Boostrix®-IPV combination vaccine.
  Interventions: Biological: Boostrix®-IPV combination vaccine
- Adults aged between 60-70 years of age (Active Comparator): Older adults from 60 up to 70 years of age determined by date of birth (dd/mm/yyyy), at the time of the first visit. Male + female, approximately equally distributed, n = 25 in each country. They will receive Boostrix®-IPV combination vaccine.
  Interventions: Biological: Boostrix®-IPV combination vaccine

INTERVENTIONS:
Biological: Boostrix®-IPV combination vaccine — A licensed aP (acellular) booster vaccine developed by GlaxoSmithKline.

SUMMARY:
This study aims to investigate the effects of aP booster vaccination in children, young adults and elderly on the (long-term) immune response to B. pertussis in three European countries with a different epidemiological background and primary vaccination schedule for pertussis.

DETAILED DESCRIPTION:
The study will be performed in three European countries (UK, Finland and the Netherlands) with a different epidemiological background for pertussis incidence and different age groups will have had different primary schedules with whole cell pertussis (wP) or aP vaccines in their first year of life. Long-term memory responses will be analysed following aP booster vaccination including a detailed assessment of antigen-specific B and T cell responses, serology assays for pertussis antigens and the effect of booster vaccination on dynamic changes in immune cell subsets and gene transcription.

There will be four cohorts of healthy volunteers:

Cohort A - children aged between 7-10 years

Cohort B - children aged between 11-15 years

Cohort C - adults aged between 20 to 34 years

Cohort D - adults aged between 60-70 years

Participants will receive one injection of reduced diphtheria toxoid, tetanus toxoid and reduced acellular pertussis vaccine (dTap)-IPV, (Boostrix® IPV, GlaxoSmithKline (GSK)) combination vaccine intramuscularly in the upper arm. Children (cohorts A and B) will be asked to donate blood four times at different time points, and young and older adults (cohorts C and D) will be asked to donate blood at set time points five times in total over the 12 months duration of the study. The time points will be:

* Timepoint 0 - day of vaccination
* Timepoint 1 - 1 day after T0 +/- 4 hours
* Timepoint 2 - 7 days after T0 +/- 1 day
* Timepoint 3 - 14 days after T0 +/- 4 days
* Timepoint 4 - 28 days after T0 +/- 4 days
* Timepoint 5 - 1 year after T0 +/- 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Normal general health
* Within the right age group for the cohort
* Received all regular vaccines for their age group according to the Dutch NIP, UK NIP or Finnish NIP; a copy of the vaccination booklet will be included in the participant's documents. If booklet is not available for cohorts A, B and C, vaccination status will be checked although, for cohort C and D this booklet might not be available due to their age;
* Provision of written informed consent
* Willing to adhere to the protocol and be available during the study period.

Exclusion Criteria:

* Present evidence of serious disease(s) within the last 3 months before inclusion requiring immunosuppressive or immune modulating medical treatment, such as systemic corticosteroids, that might interfere with the results of the study;
* Chronic infection
* Known or suspected immune deficiency;
* History of any neurologic disorder, including epilepsy;
* Previous administration of serum products (including immunoglobulins) within 6 months before vaccination and blood sampling;
* Known and/or suspected allergy to any of the vaccine components (by medical history);
* Occurrence of a serious adverse events (SAEs) after primary DTwP-IPV vaccination, DTaP-IPV vaccination or any other vaccination (by medical history);
* Vaccination with any other pertussis vaccine other than those described in the inclusion criteria (i.e. only according to NIP)
* Vaccination with any other DT-IPV vaccine in the last 5 years, a DT-IPV vaccination according to NIP in cohort B is not an exclusion criterion;
* Children between 8 and 10 years of age eligible for cohort A in the Netherlands who have already received the diphtheria and tetanus toxoid vaccine (DT)-IPV booster vaccination according to Dutch NIP around 9 years of age;
* Mixed wP and aP priming within a participant, cohort B;
* Pregnancy. Detailed considerations for this exclusion criteria in section 4.6.

Temporary exclusion criteria

* If a participant has a severe acute (infectious) illness or fever (>38°C) within 14 days prior to T0, participation will be postponed or cancelled. In case the participant has fever within 2 days before sampling at T4 or T5, the appointment will be postponed for 4 days, if possible.
* Antibiotic use within 14 days of enrolment.
* Any vaccination within a month before enrolment.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pertussis toxin-specific IgG antibody levels to 28 days after vaccination | 28 days

SECONDARY OUTCOMES:
Amount of pertussis toxin (PT) specific IgG antibody one year after vaccination with Boostrix-IPV | 1 year
Change from baseline in pertussis toxin (PT) specific IgG-subclasses and avidity levels to 28 days and 1 year after vaccination with Boostrix-IPV | 28 days and 1 year
Change from baseline of antigen-specific IgG antibody levels against other pertussis vaccine antigens (such as FHA) and non-pertussis vaccine antigens (such as diptheria and tetanus toxoid) to 28 days and 1 year after vaccination with Boostrix-IPV | 28 days and 1 year
Change from baseline of functional pertussis-specific antibody levels to 28 days and 1 year after vaccination with Boostrix-IPV | 28 days and 1 year
Change from baseline of B cell responses against Bordetella pertussis vaccine proteins after vaccination with Boostrix-IPV | 7 days, 28 days and 1 year
  Antigen-specific memory B cell responses against B-pertussis vaccine proteins
Change from baseline of pertussis antigen-specific T helper responses to 14 days, 28 days and 1 year after vaccination with Boostrix-IPV | 14 days, 28 days and 1 year
  To describe the effect on an aP booster on the specific T cell immune response in different age groups that have been initially vaccinated with either a whole cell or acellular vaccine
Identify markers in biological samples collected in the Biobank (library of samples) that show changes in immunity to pertussis | 1 year although samples will be stored up to 10 years
  Use of novel exploratory immunoassays on stored samples to identify biomarkers or lasting memory or waning immunity to pertussis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marlies van Houten, Principal Investigator — Spaarne Hospital, Hoofddorp; Prof. dr. Jussi Mertsola, Principal Investigator — Turku University Hospital; Dr Dominic Kelly, Principal Investigator — University of Oxford
Locations (3):
- University of Turku, Turku, Finland
- Centre for Infectious Disease Control, National Institute for Public Health and the Environment (RIVM), Bilthoven, Netherlands
- Centre for Clinical Vaccinology & Tropical Medicine (CCVTM), Oxford, Oxfordshire, United Kingdom